CLINICAL TRIAL: NCT01930513
Title: Exercise Capacity and Daily Physical Activity in Obese Subjects With Treated Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Respirologist, West Park Healthcare Centre
Other Study IDs: RG2010OSA
Record Dates: First submitted 2013-07-15; First posted 2013-08-29 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Obstructive Sleep Apnea; Obesity
Keywords: Obesity; Obstructive Sleep Apnea; Exercise; Walking tests; Cardiopulmonary exercise tests; Physical activity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Obesity is very common worldwide and breathing problems at night (obstructive sleep apnea, OSA) are common in obesity. Despite the best treatment, obesity and OSA are linked to early death from heart problems. They are also associated with lower levels of physical activity. Exercise strategies for weight loss, increasing physical activity and improving fitness are needed for obesity. In Obese individuals with OSA

1. The investigators will compare corridor walking tests compared to laboratory exercise tests. The null hypothesis is that the peak oxygen uptake achieved and the cardiopulmonary response during both the six-minute walk test and Incremental Shuttle Walk Test would not be different from that observed during an Incremental Treadmill Test.
2. The investigators will investigate whether cycling or walking uses more calories for the same intensity. We hypothesise that cycling (weight supported) will be endured for long.
3. The investigators will compare commonly used exercise tests with levels of daily physical activity.

The information from these three projects will help us set up the optimal exercise program for obese individuals.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive Sleep Apnea
* Obesity BMI>30
* Controlled on Continuous Positive Airway Pressure for three months

Exclusion Criteria:

* cardiac co-morbidity e.g ischaemic heart disease, chronic heart failure, valvular heart disease
* pulmonary co-morbidity
* neurological condition limiting the ability to perform walking or cycling
* orthopaedic condition limiting the ability to perform walking or cycling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obstructive Sleep Apnea
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake (Peak VO2) measured at the end of the Incremental Shuttle Walk Test (ISWT) | All outcome measures will be performed within four weeks of each other
  Two Incremental Shuttle Walk tests will be performed within two hours on the same day with expired gas analysis measured by a portable gas analyser. An ISWT is conducted over a 10m course and the speed is externally paced and increases each minute. The participant is asked to continue until they are either too breathless or too tired to continue.

SECONDARY OUTCOMES:
Six minute walk test (6MWT) | Four weeks
  The 6MWT will be performed over a 30 m level, straight course within an enclosed corridor. The test protocol described by the American Thoracic Society will be modified to include standardized encouragement every 15 seconds to recommence walking if the participant chooses to rest during the test. Participants will be familiarized with the test prior to participating in the study and, therefore, only one test will be performed.
Incremental Treadmill Test (ITM) | Four weeks
  A maximal treadmill test will be performed once with expired gas analysis.
Incremental cycle test (ICE) | Four weeks
  A maximal symptom limited cardio-pulmonary exercise test on a cycle ergometer.
Endurance cycle ergometer | Four weeks
  Two endurance cycle tests will performed at 60% and 80% of the maximal peak oxygen obtained on either the ICE or ITM
Endurance treadmill test | Four weeks
  Constant speed endurance treadmill test will be performed at 60% and 80% of the peak oxygen uptake achieved on either the ITM or ICE to symptom limitation
Daily physical activity | Four weeks
  A sensewear armband will be worn for 7 days and only taken off for showering/bathing.

CONTACTS AND LOCATIONS:
Overall Officials: Roger S Goldstein, MBChB, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Evans RA, Dolmage TE, Robles PG, Goldstein RS, Brooks D. Do field walking tests produce similar cardiopulmonary demands to an incremental treadmill test in obese individuals with treated OSA? Chest. 2014 Jul;146(1):81-87. doi: 10.1378/chest.13-2060. PMID 24577643